CLINICAL TRIAL: NCT04936698
Title: The Prevalence and Risk Factors for Thyroid Dysfunction in Pregnant Women in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202100365B0
Record Dates: First submitted 2021-06-17; First posted 2021-06-23 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-06

CONDITIONS: Thyroid Disease Pregnancy
MeSH Terms: interventions — Tablets; Thyroxine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hyperthyroidism: Elevated fT4, low TSH
  Interventions: Drug: PTU 50 MG Oral Tablet
- Hypothyroidism: Elevated TSH, low fT4
  Interventions: Drug: Levothyroxin
- Euthyroid: Normal TSH/fT4 level

INTERVENTIONS:
Drug: PTU 50 MG Oral Tablet — to treat if the patient has hyperthyroidism
  Groups: Hyperthyroidism
Drug: Levothyroxin — to treat if the patient has hypothyroidism
  Groups: Hypothyroidism

SUMMARY:
The investigators' aim is to enroll around 2000 patients from Taipei, Keelung, Linkou, Chiayi and Kaohsiung CGMH. All participants will receive universal thyroid function screening at 1st trimester, and those who was found to have hyperthyroidism or hypothyroidism will be referred to Endocrine department for further treatment. All participants will be followed at outpatient clinic, and their obstetric visit finding will be recorded. The maternal and neonatal outcomes will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at first trimester (< 14 weeks of gestational age)

Exclusion Criteria:

* None

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women at their first trimester of pregnancy may be enrolled.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
The prevalence thyroid dysfunction | 40 weeks
  Hypothyroidism: defined as serum TSH > 2.5U/mL and decreased fT4*; Hyperthyroidism: defined as fT4 > normal range* and TSH undetectable
  * Serum free T4 range varies according to trimesters.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
The decision will be made once the study is completed.